CLINICAL TRIAL: NCT06131710
Title: Effects of Proximal Strengthening Exercises on Pain and Function in Patellofemoral Pain Syndrome Among Basketball Players
Brief Title: Effects of Proximal Strengthening Exercises in Patellofemoral Pain Syndrome Among Basketball Players
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/23/0430
Record Dates: First submitted 2023-11-09; First posted 2023-11-14 (Actual); Last update posted 2024-01-30 (Actual); Status verified 2024-01

CONDITIONS: Patellofemoral Syndrome
Keywords: Clamshell; Isolated exercise; Pain; Patellofemoral syndrome; Squat
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Isolated Strengthening Exercises (Experimental): Isolated strengthening exercises refers to set of exercises that are used to treat a specific part of body. In our study, isolated strengthening exercises including 10 repetition of 3 sets of legs extensions,10 repetition of 3 sets squats and 10 repetition of 3 sets lunges are used. These exercises aim to improve the pain and range of motion of knee by acting on quadriceps.
  Interventions: Other: Isolated Strengthening Exercises
- Combined Strengthening Exercises (Experimental): The Combined strengthening group will perform the same isolated strengthening exercises, but with the addition of proximal strengthening exercises for the hip and core muscles. These exercises include 10 repetitions of bridging(3 sets), 10 repetitions of clamshells(2 sets), 10 repetition of 3 sets of legs extensions,10 repetition of 3 sets squats,10 repetition of 3 sets lunges and 10 repetitions of planks(2 sets).
  Interventions: Other: Isolated Strengthening Exercises; Other: Combined Strengthening Exercises

INTERVENTIONS:
Other: Isolated Strengthening Exercises — Isolated strengthening exercises can be beneficial for individuals with Patellofemoral Pain Syndrome (PFPS) to help address muscle imbalances and alleviate pain.
Other: Combined Strengthening Exercises — Combined strengthening exercises for Patellofemoral Pain Syndrome (PFPS) typically include a mix of quadriceps strengthening exercises, hip strengthening exercises, and core stability exercises. The goal is to address muscle imbalances and improve the overall stability of the knee joint.
  Arms: Combined Strengthening Exercises

SUMMARY:
This research study aims to compare the effectiveness of two different exercise approaches in treating Patellofemoral Pain Syndrome (PFPS) in basketball players. It employs a randomized clinical trial with 32 participants aged 18-40 diagnosed with PFPS. The participants are divided into two groups: Isolated Strengthening Exercises (ISE) and Combined Strengthening Exercises (CSE). The ISE group focuses solely on quadriceps strengthening exercises, while the CSE group incorporates both quadriceps and proximal strengthening exercises for the hip and core muscles. Outcome measures include pain levels, functionality, and physical performance assessments recorded at baseline and after 6 weeks. Statistical analysis using independent t-tests in SPSS will determine which approach is more effective. This study seeks to provide evidence on whether the combination of proximal strengthening exercises enhances the reduction of pain and improvement in functionality for basketball players with PFPS, compared to isolated strengthening exercises alone.

DETAILED DESCRIPTION:
Patellofemoral Pain Syndrome (PFPS) is a common knee condition that affects basketball players and can lead to significant pain and functional limitations. The syndrome involves pain around or behind the patella (kneecap) due to malalignment and abnormal tracking of the patella within the femoral groove. Isolated strengthening exercises targeting the quadriceps have been widely recommended as a treatment approach for PFPS. However, recent research suggests that incorporating proximal strengthening exercises, focusing on the hip and core muscles, may enhance treatment outcomes. This study aims to investigate the comparative effectiveness of isolated strengthening exercises alone versus combined with proximal strengthening exercises in reducing pain and improving functionality in basketball players with PFPS. This research will employ a randomized clinical trial design to assess the impact of different strengthening exercise protocols on pain and functionality among basketball players diagnosed with PFPS. A sample of 32 basketball players aged 18-40 years, diagnosed with PFPS by a qualified orthopedic specialist and physiotherapists will be recruited for the study. Participants will be randomly assigned into two groups: The Isolated Strengthening Exercises (ISE) group and the Combined Strengthening Exercises (CSE) group, which includes both isolated and proximal strengthening exercises. The ISE group will follow a structured program consisting of isolated strengthening exercises targeting the quadriceps, focusing on exercises such as leg extensions, squats, and lunges. The CSE group will perform the same isolated strengthening exercises but with the addition of proximal strengthening exercises for the hip and core muscles, including exercises such as hip abduction, clamshells, and planks. Outcome measures, including pain levels using NPRS, functionality using the KOOS-PF, Step-down test, single leg squat Hop test, and range of motion assessments, will be recorded at baseline after 6 weeks. Statistical analysis, including independent t-tests, will be performed to compare the outcomes between the ISE and CSE groups using SPSS version 26.0.

ELIGIBILITY:
Inclusion criteria:

* Professional male basketball players of the age group 18-40 years
* Practicing players of basketball (3-5 times a week)
* Players who experience pain around Patella
* Pain severity between 3 and 10 during stair descending test for PFPS
* Positive diagnostic patellofemoral syndrome maneuvers including Shrug test, Grind test and Perkins test

Exclusion criteria:

* Past surgery of affected leg
* Systemic illness (diabetes, systemic lupus erythematosus)
* Individuals havening significant knee pathologies such as ACL tear, Meniscal tear
* Referred pain originating from other points of body
* Knee deformities or signs of knee OA in knee x-ray

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-05-05 (Actual); Primary Completion 2024-02-05 (Estimated); Study Completion 2024-02-05 (Estimated)

PRIMARY OUTCOMES:
Numeric pain rating scale | 6 weeks
  The Numeric pain rating scale is a self-reported, or clinician-administered, measurement tool consisting of a numerical point scale with extreme anchors of no pain to extreme pain. The scale is typically set up on a horizontal or vertical line, ranges most commonly from 0-10 or 0-100, and can be administered in written or verbal form. The 0 on scale shows no pain, 1-4 shows mild pain, 5 and 6 shows moderate pain and 7-10 shows severe pain.
Knee Injury and Osteoarthritis outcome score for Patellofemoral injury | 6 weeks
  Knee Injury and Osteoarthritis Outcome Score Patellofemoral is one subjective type of questionnaire developed as an extension with the aim of estimating the immediate and long-term symptoms and function among people with Patellofemoral pain syndrome. Higher scores show pain severity whereas lower score shows mild or no pain.
Single-legged hop tests | 6 weeks
  Single-legged hop tests are functional tests that have been used to identify individuals who can regain dynamic knee stability after an ACL injury.

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Asrar Yousaf, PhD, Principal Investigator — Riphah International University
Locations (1):
- Physio wellness centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mostafaee N, Pashaei-Marandi M, Negahban H, Pirayeh N, Saki Malehi A, Ebrahimzadeh MH. Examining the diagnostic accuracy of common physical examination and functional tests in the diagnosis of patellofemoral pain syndrome among patients with anterior knee pain. Physiother Theory Pract. 2024 Apr;40(4):843-855. doi: 10.1080/09593985.2022.2158053. Epub 2022 Dec 19. PMID 36537113
- [Background] You S, Shen Y, Liu Q, Cicchella A. Patellofemoral Pain, Q-Angle, and Performance in Female Chinese Collegiate Soccer Players. Medicina (Kaunas). 2023 Mar 16;59(3):589. doi: 10.3390/medicina59030589. PMID 36984590